CLINICAL TRIAL: NCT01931904
Title: Observational Study of Ocular Blood Flow Pre- and Post- Glaucoma Surgery Using Functional and Structural Optical Coherence Tomography
Brief Title: Eye Pressure Lowering Surgery
Acronym: IOP
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Aiyin Chen, MD, Associate Professor of Ophthalmology, Glaucoma Services Director, Oregon Health and Science University
Other Study IDs: IRB000009745; 1R01EY023285 (NIH)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
Keywords: IOP; Glaucoma; Trabeculectomy
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trabeculectomy or Tube Shunt Patients: 46 glaucoma patients undergoing trabeculectomy or tube shunt surgery to lower IOP

SUMMARY:
The purpose of this study is to determine if lowering the pressure inside the eye improves blood flow to the eye.

DETAILED DESCRIPTION:
Using high-speed ocular coherence tomography (OCT) systems, we have developed new methods to image and measure optic nerve head (ONH) and retinal blood flow. Preliminary results have shown that visual field (VF) loss is more highly correlated with retinal blood flow as measured by OCT than any neural structure measured by OCT or other imaging modality. Accordingly, the goal of the proposed project is to improve the diagnostic and prognostic evaluation of glaucoma by further developing novel functional OCT measurements using ultrahigh-speed (70-100 kHz) OCT technology.

Retinal blood flow, ONH circulation, optic disc rim volume, peripapillary nerve fiber layer volume, and macular ganglion cell complex volume are all pieces of the same glaucoma puzzle. This project will develop novel imaging methods that allow us to look at the whole picture using one tool - ultrahigh-speed OCT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with perimetric open angle glaucoma or chronic angle closure glaucoma.
* Subjects scheduled to undergo trabeculectomy or tube shunt surgery

Exclusion Criteria:

* Best-corrected visual acuity less than 20/40
* Age < 18 or >85 years
* Refractive error of > +3.00 D or < -7.00 D
* Previous vision correction surgery such as Laser-Assisted in situ Keratomileusis (LASIK) or Photorefractive Keratectomy (PRK)
* Previous intraocular surgery except for uncomplicated cataract extraction with posterior chamber intraocular lens implantation
* Diabetic retinopathy
* History of heart failure, myocardial infarction, transient ischemic attack or stroke
* Other diseases that may cause VF loss or optic disc abnormalities
* Inability to clinically view or photograph the optic discs due to media opacity or poorly dilating pupil
* Inability to perform reliably on automated VF testing
* Life-threatening or debilitating illness making it unlikely patient will successfully complete the study.
* Refusal of informed consent or of commitment to the full length of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will measure blood flow changes in 46 glaucoma patients undergoing trabeculectomy or shunt surgery to lower IOP.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Effects of Intraocular Pressure (IOP) Reduction on Ocular Perfusion | Subjects will be evaluated on enrollment (pre-operatively) and at post-operative visits ( 3, 6, 12, 18, and 24-months post-op).
  To determine if IOP reduction improves ocular perfusion. Change in IOP reduction will be measured in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Aiyin Chen, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

REFERENCES:
- See also: Related Info — http://coollab.net